CLINICAL TRIAL: NCT03859297
Title: Developing Rumination-focused Treatment to Reduce Risk for Depression Recurrence (RDR) in Adolescence
Brief Title: Mechanisms of Rumination Change in Adolescent Depression
Acronym: RuMeChange
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Exeter (Other); National Institute of Mental Health (NIMH) (NIH); University of Utah (Other); Nationwide Children's Hospital (Other); Utah Center for Evidence Based Treatment (Unknown)
Responsible Party: Principal Investigator, Scott Langenecker, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB_00113733; R61MH116080 (NIH)
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder; Mood Disorders
Keywords: rumination; depression; brain imaging; cognitive behavioral therapy; rumination focused cognitive behavioral therapy; default mode network; rumination induction
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Rumination Syndrome; Depression

STUDY DESIGN:
Intervention Model Description: First two years. randomization to either rumination-focused cognitive behavioral therapy (RF-CBT) or Assessment only (AO) for a 10 week intervention period.
  Last three years. randomization to either rumination-focused cognitive behavioral therapy (RF-CBT) or Relaxation therapy (RelaxT) for a 10 week intervention period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rumination-Focused CBT (Experimental): RF-CBT is a manual-based treatment for prevention of depression, includes focus on ruminations, mental habits, concreteness training, and mindfulness.
  Interventions: Behavioral: Rumination-Focused CBT
- Treatment as Usual (No Intervention): Participants are allowed to continue any therapy outside of the treatment study.
- Relaxation-based therapy (Active Comparator): RelaxT includes an active comparison treatment that can be used to monitor and modify physiological responses to stress
  Interventions: Behavioral: Relaxation-based Therapy

INTERVENTIONS:
Behavioral: Rumination-Focused CBT — RF-CBT targets rumination and other maladaptive forms of emotion regulation such as suppression and avoidance and provides skills training in effectively coping with rumination. RF-CBT specifically targets rumination through psychoeducation, adopting a functional analytic approach to the learned habitual behavior of rumination, and a focus on shifting process style. The adolescent is taught to notice triggers to ruminate as well as the consequences of rumination and to shift into practicing a more adaptive strategy such as an attention training exercise, behavioral activation, thinking in a concrete way, or active problem-solving. RF-CBT directly teaches adolescents to recognize rumination or "when the participant gets stuck in their head" and to notice the influence this has on their mood.
  Arms: Rumination-Focused CBT
Behavioral: Relaxation-based Therapy — Sessions will include progressive muscle relaxation, simple breathing techniques, and guided imagery that focus on bodily and somatic relaxation. Adolescents randomized to Relaxation Therapy (RelaxT) will also receive exercises to do as homework in between sessions, parallel to the RF-CBT group.
  Arms: Relaxation-based therapy

SUMMARY:
This study will evaluate whether a newer treatment, rumination-focused cognitive behavioral treatment, which includes mindfulness and can be used to reduce ruminative habits, change ways in which key brain regions interact with each other (e.g.., often called connectivity), and whether these changes in habits and brain connectivity can reduce the risk for recurrence of depression in the next two years.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a disease that has it's onset in childhood and early adolescence for many. Treatments in adolescence tend to be acute and short-term. Unfortunately, between half and three quarters of adolescents who have a first episode of MDD will go to have a second episode within the next two years. Studies in adults suggest that maintenance treatments or preventative treatments can lower these risks and delay or stop recurrences.

The present study will use a preventative strategy, rumination-focused CBT (RF-CBT) to delay or stop the onset of another MD episode for at least two years.

For the first 2 years of the study, adolescents with a history of MDD who are currently well will be randomly selected for either treatment with RF-CBT or just treatment as usual in the first two years of the study.

In the last 3 years of the study, these adolescents will be randomized to either RF-CBT or Relaxation Therapy above and beyond TAU (Treatment as Usual). Brain, cognitive, and self-report measurements are collected before during and after the intervention to evaluate what brain and rumination changes occur, and which adolescents benefit the most from the treatment.

What will happen.

1. The Investigators determine if the child is eligible (see criteria below for 14-17 year olds with history of MDD.
2. The Investigators complete pre-intervention assessments with the child that include

   1. brain imaging
   2. tests of cognitive skills and emotion processing, including rumination
   3. questionnaires about how the adolescent thinks and responds to situations, similar questionnaires in at least one parent/guardian
   4. measurement of sleep using a handheld wristwatch (called an actigraph - optional).
3. randomization (chance assignment) in years 1-2 to either rumination focused cognitive behavioral therapy (RF-CBT) or assessment only for a 10-14 session intervention. Treatment as usual continues for all adolescents. In years 3-5, chance assignment is to RF-CBT or Relaxation Therapy.
4. repeat assessments after the intervention period. The cognitive skills and emotion processing are also assessed during the middle of the intervention period.

   1. brain imaging
   2. tests of cognitive skills and emotion processing, including rumination
   3. questionnaires about how the adolescent thinks and responds to situations, similar questionnaires in at least one parent/guardian
   4. measurement of sleep using a handheld wristwatch (called an actigraph - optional).
5. follow-up assessments to determine any changes, recurrence of depression, new treatments for the next two years.

   1. questionnaires
   2. interviews

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of Major Depressive Disorder (full or partial remission for at least two weeks) according to Diagnostic and Statistical Manual (DSM-V) criteria confirmed by the Kiddie Schedule for affective disorders (KSADSPL). Partial remission is defined as not meeting full DSM-V criteria for MDD.
* RRS score above the age and sex specific mean, T > 50).
* 14-17 years of age at enrollment (accounting for 2 year follow-up),
* Postpubertal (Petersen Pubertal Developmental Scale)
* Youth assent and parent consent
* Intellectual Quotient (IQ) > 75, determined by Wechsler Abbreviated Scale of Intelligence (WASI)

Exclusion Criteria:

* Endorsement of suicidality with plan or intent (assessed via KSADSPL and Children's Depression Rating Scale (CDRS-R) clinical interviews. Current or past (within previous three months) plan or intent is exclusionary.
* Lifetime history of conduct disorder, autism, any psychotic disorder (or episode unexplained by other known medical causes), or bipolar disorder. Eating disorder or alcohol/substance abuse within the previous 6 months. (Lifetime history of an anxiety disorder, disruptive mood dysregulation disorder or oppositional defiant disorder, Attention Deficit Hyperactivity Disorder (ADHD) will not be exclusionary).
* Current treatment with RF-CBT, Cognitive Behavioral Therapy (CBT), or variants thereof, or in the last 2 years. Likewise, detail oriented therapy beyond supportive therapy (e.g., homework, cognitive restructuring), in same time window (ability to recall elements of structured therapies with CBT focus).
* Metal braces or retainers, tattoos with metal, or clothing with metal fibers.
* Claustrophobia
* Current pregnancy - Parents will be asked this information at the phone screen. At the clinic eligibility visit, female participants will be asked about sexual activity in a private room separate from their parents using the pregnancy script/screen that the investigators have created. This script details that if a female is ineligible due to pregnancy or inadequate birth control, this information will not be disclosed to her parent(s). Participants who are sexually active will be asked about birth control method. Abstinence will be considered an approved form of contraception.
* Psychotropic medication outside of antidepressants such as mood stabilizers and antipsychotics will be exclusionary. Participants may have a history of current, stable antidepressant medication use, with no changes in dose for the past four weeks, no change in specific medication for six weeks.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — all gender representations are allowed.
Enrollment: 183 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-04-14 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Rumination Responsiveness Scale (RRS) | ~14-22 weeks
  RRS is a scale developed by Dr. Susan Nolan-Hoeksema that is used to determine pre-post reductions in rumination after RF-CBT.
  The RRS is the Rumination Responsiveness Scale. Scores range from a low of 22 to a high of 88 on the 232 item scale. Higher scores indicate more difficulties with rumination. Higher rumination has been reported in a number of samples of both active and remitted MDD.
  The outcome is a reliable change index decline of at least 1/2 standard deviation in the RF-CBT group relative to the AO and RelaxT arms.
  In our preliminary study, the RRS declined from 52.88 to 43 (Jacobs et al., 2016). An age matched control group had a mean score of 30.4 (7.1), Burkhouse et al., 2016.
Resting state functional magnetic resonance imaging (fMRI) connectivity of Default mode network to cognitive control network. | ~14-22 weeks
  Using seed based approaches with the posterior cingulate gyrus and medial prefrontal cortex, the investigators will evaluate if RF-CBT and not AO or RelaxT, results in decreases in rs-fMRI connectivity to cognitive control network nodes, particularly right inferior frontal and temporal gyri.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Langenecker, Ph.D., Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data relevant to the clinical trial and primary R61/R33 targets will be release biannually per requirements of the NIH policy, the request for application (RFA) and consistent with HIPAA and Institutional Review Board (IRB) approval at the University of Utah and the University of Exeter. In addition to the data for the clinical trial specifically, demographic and clinical information will be included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared in line with Resource Sharing guidelines for this specific RFA
Access Criteria: Available to researchers, after appropriate data sharing agreements have been made with the University of Utah.

REFERENCES:
- [Background] Watkins ER, Mullan E, Wingrove J, Rimes K, Steiner H, Bathurst N, Eastman R, Scott J. Rumination-focused cognitive-behavioural therapy for residual depression: phase II randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):317-22. doi: 10.1192/bjp.bp.110.090282. Epub 2011 Jul 21. PMID 21778171
- [Background] Burkhouse KL, Jacobs RH, Peters AT, Ajilore O, Watkins ER, Langenecker SA. Neural correlates of rumination in adolescents with remitted major depressive disorder and healthy controls. Cogn Affect Behav Neurosci. 2017 Apr;17(2):394-405. doi: 10.3758/s13415-016-0486-4. PMID 27921216
- [Background] Jacobs RH, Watkins ER, Peters AT, Feldhaus CG, Barba A, Carbray J, Langenecker SA. Targeting Ruminative Thinking in Adolescents at Risk for Depressive Relapse: Rumination-Focused Cognitive Behavior Therapy in a Pilot Randomized Controlled Trial with Resting State fMRI. PLoS One. 2016 Nov 23;11(11):e0163952. doi: 10.1371/journal.pone.0163952. eCollection 2016. PMID 27880789
- [Background] Hvenegaard M, Watkins ER, Poulsen S, Rosenberg NK, Gondan M, Grafton B, Austin SF, Howard H, Moeller SB. Rumination-focused cognitive behaviour therapy vs. cognitive behaviour therapy for depression: study protocol for a randomised controlled superiority trial. Trials. 2015 Aug 11;16:344. doi: 10.1186/s13063-015-0875-y. PMID 26260780
- [Background] Watkins ER, Nolen-Hoeksema S. A habit-goal framework of depressive rumination. J Abnorm Psychol. 2014 Feb;123(1):24-34. doi: 10.1037/a0035540. PMID 24661156
- [Background] McEvoy PM, Watson H, Watkins ER, Nathan P. The relationship between worry, rumination, and comorbidity: evidence for repetitive negative thinking as a transdiagnostic construct. J Affect Disord. 2013 Oct;151(1):313-20. doi: 10.1016/j.jad.2013.06.014. Epub 2013 Jul 16. PMID 23866301
- [Background] Dillahunt AK, Feldman DA, Thomas LR, Farstead BW, Frandsen SB, Lee S, Pazdera M, Galloway J, Bessette KL, Roberts H, Crowell SE, Watkins ER, Langenecker SA, Westlund Schreiner M. Self-Injury in Adolescence Is Associated with Greater Behavioral Risk Avoidance, Not Risk-Taking. J Clin Med. 2022 Feb 26;11(5):1288. doi: 10.3390/jcm11051288. PMID 35268378
- [Derived] Roberts H, Jacobs RH, Bessette KL, Crowell SE, Westlund-Schreiner M, Thomas L, Easter RE, Pocius SL, Dillahunt A, Frandsen S, Schubert B, Farstead B, Kerig P, Welsh RC, Jago D, Langenecker SA, Watkins ER. Mechanisms of rumination change in adolescent depression (RuMeChange): study protocol for a randomised controlled trial of rumination-focused cognitive behavioural therapy to reduce ruminative habit and risk of depressive relapse in high-ruminating adolescents. BMC Psychiatry. 2021 Apr 23;21(1):206. doi: 10.1186/s12888-021-03193-3. PMID 33892684